CLINICAL TRIAL: NCT03569540
Title: Glibenclamide in Aneurysmatic Subarachnoid Hemorrhage: A Prospective and Randomized Study
Brief Title: Glibenclamide in Aneurysmatic Subarachnoid Hemorrhage
Acronym: GASH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 55947016.2.0000.0068
Record Dates: First submitted 2018-05-17; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-01

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
Keywords: Subarachnoid hemorrhage; Glibenclamide
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Glyburide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treated Patients (Experimental): Patients who will receive Glibenclamide 05mg daily for 21 days, orally or by nasogastric tube.
  Interventions: Drug: Glibenclamide
- Control Group (Placebo Comparator): Patients who will receive amylum 05mg daily for 21 days, orally or by nasogastric tube.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Glibenclamide — Placebo-controlled; Double blind test
  Arms: Treated Patients
Other: Placebo — Amylum
  Arms: Control Group

SUMMARY:
A randomized, double-blind and prospective trial meant to evaluate the use of Glibenclamide on acute aneurysmatic subarachnoid hemorrhage. Patients will allocated randomly in two groups, one for 05 mg daily intake of glibenclamide for 21 days and another for control with placebo. General clinical data and late cognitive status will be accessed in both groups.

DETAILED DESCRIPTION:
GASH is a double blind, prospective and randomized clinical trial centered on the University of Sao Paulo General Hospital. Patients will be recruited from neurological/neurosurgical intensive care units. Appropriate ethics and regulatory approvals will be sought for all subjects, according to the International Conference on Harmonization guidelines for good clinical practice (ICH GCP). Investigators will obtain informed written consent from all patients or their legal representative. Recruitment will take place between 2018 and 2019.

Patients will be randomly assigned (1:1) to receive either glibenclamide 5mg or placebo. Coded boxes containing either 21 similar tablets of glibenclamide 5mg or placebo will be assigned a number. A computer-generated randomization code will be used to randomize patients by blocks of ten (five glibenclamide, five placebo). Each box will be identified by a code number specific and subsequently selected for distribution in ascending numerical order. Patients will start treatment as soon as possible within 96 h of the ictus, with a daily dose till the 21° day after the bleed. Trial medication consisted of one tablet a day, given orally or via a nasogastric tube. Aneurysm treatment, either by microsurgery or embolization, will be performed as soon as possible, according with the standard of care for the recruiting center. Nimodipine 60mg, every four hours, will be started on admission and continued till the 21° day after the ictus, in all patients as standard of care.

Patient's demographics, medical history and relevant investigation results will be collected. The severity of the hemorrhage will be clinically assessed by World Federation of Neurosurgical Societies grading scale and radiologically using the modified Fischer scale. At 6 months of follow up patients will be interviewed with modified Rankin scale (mRS) questionnaire (a scale that measures degree of incapacity/ dependence and mortality after neurological events) by a nurse or a physician with no knowledge of treatment allocation. Psychologists will evaluate quality of life and cognitive performance using the "short-form health survey questionnaire" (SF-36) and neuropsychological tests. The main hypothesis is that, once compared with standard of care, glibenclamide 5mg will provide better clinical outcome and additionally will decrease mortality and improve quality of life and cognitive performance after 6 months.

Sample size: It was estimated the sample size of 50 randomized patients to give 90% power at the 5% significance level (two-sided) to detect a treatment effect equivalent to an absolute increase of 7% in the proportion of patients with a favorable outcome (30-day mortality rate after subarachnoid hemorrhage approaches 50% and 25% of survivors present some degree of neurological morbidity25). This calculation was based on an ordinal analysis of the 6-month mRS (the primary outcome) assuming that the treatment effect follows a proportional odds model.

ELIGIBILITY:
Inclusion Criteria:

* Radiological confirmatory evidence of an aneurysmal subarachnoid hemorrhage (by digital subtraction angiography, CT angiography, or magnetic resonance angiography)
* Presentation less than 96 h from ictus

Exclusion Criteria:

* Patients taking glibenclamide therapy at presentation
* Pregnancy
* Hunt & Hess V
* Known renal or hepatic impairment
* Patient not fully independent before bleed,
* Strong suspicion of drug or alcohol misuse
* Patient taking warfarin-type drugs
* Suspected additional life-threatening disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-07-03 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (early) | To be measured on the 21th day of medication/control, when happens the end of intervention
  Evaluate patients life quality and morbidity, from 1 to 6 ('no symptoms' to 'Death')
Short-Form Healthy Survey Questionnaire (SF-36) | To be executed 6 months after the end of intervention
  Cognitive assessment and quality of Life measured by 11 questions that leads to a quantification scale called Raw Scale (RS). The RS identify 8 domains with a calculable score from 0 (worst) to 100 (best): Functional capacity; Limitation by physical aspects; Pain; General health; Vitality; Social aspects; Emotional aspects and Mental health.
Modified Rankin Scale (late) | To be measured 6 months after the end of intervention and compared with the early result
  Evaluate patients life quality and morbidity, from 1 to 6 ('no symptoms' to 'Death')

CONTACTS AND LOCATIONS:
Overall Officials: Isabela Windlin, Study Chair — Neuropsicology
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] da Costa BBS, Windlin IC, Koterba E, Yamaki VN, Rabelo NN, Solla DJF, Teixeira MJ, Figueiredo EG. Glibenclamide in aneurysmatic subarachnoid hemorrhage (GASH): study protocol for a randomized controlled trial. Trials. 2019 Jul 9;20(1):413. doi: 10.1186/s13063-019-3517-y. PMID 31288831